CLINICAL TRIAL: NCT01001650
Title: A Phase 1/2a Trial of the PfSPZ Vaccine Administered Subcutaneously or Intradermally to Malaria-Naïve Adult Volunteers
Brief Title: Clinical Trial of the PfSPZ Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Sanaria.2008.001; NMRC.2008.0004; NNMC: 2008.0071; CVD-UMB Site: H-30076; Malaria CVD 18000; WRAIR DHSP: #1487; HRPO: A-14947; PATH MVI: #PfSPZ001
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Plasmodium Falciparum
Keywords: Malaria Vaccine; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 4 doses of 7,500 PfSPZ/immunization.
  Interventions: Biological: Plasmodium falciparum Sporozoite (strain NF-54; Anopheles stephensi mosquitoes) Vaccine, Live, Inactivated (gamma irradiation)
- Group 2 (Experimental): 4 doses of 30,000 PfSPZ/immunization
  Interventions: Biological: Plasmodium falciparum Sporozoite (strain NF-54; Anopheles stephensi mosquitoes) Vaccine, Live, Inactivated (gamma irradiation)
- Group 3 (Experimental): 4 doses of 135,000 PfSPZ/immunization
  Interventions: Biological: Plasmodium falciparum Sporozoite (strain NF-54; Anopheles stephensi mosquitoes) Vaccine, Live, Inactivated (gamma irradiation)
- Group 4 (Experimental): 4 or 6 doses of 135,000 PfSPZ/immunization.
  Interventions: Biological: Plasmodium falciparum Sporozoite (strain NF-54; Anopheles stephensi mosquitoes) Vaccine, Live, Inactivated (gamma irradiation)

INTERVENTIONS:
Biological: Plasmodium falciparum Sporozoite (strain NF-54; Anopheles stephensi mosquitoes) Vaccine, Live, Inactivated (gamma irradiation) — Group 1: 4 doses of 7,500 PfSPZ/immunization,
  Group 2: 4 doses of 30,000 PfSPZ/immunization,
  Group 3: 4 doses of 135,000 PfSPZ/immunization, and
  Group 4: 4 or 6 doses of 135,000 PfSPZ/immunization.
  If > 80% protective efficacy is not achieved in Groups 1, 2, or 3, volunteers in Group 4 will receive a fifth and sixth dose.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of a non-replicating, metabolically active Plasmodium falciparum sporozoite (PfSPZ) vaccine in malaria-naïve healthy volunteers following multiple-dose subcutaneous (SC) or intradermal (ID) administration.

In addition, the investigators wish to evaluate PfSPZ vaccine-mediated protection against P. falciparum challenge in the following 4 groups (see below) and compare protective efficacy of the PfSPZ vaccine when given by SC v ID administration in all these groups:

* Group 1: 4 doses of 7,500 PfSPZ/immunization,
* Group 2: 4 doses of 30,000 PfSPZ/immunization,
* Group 3: 4 doses of 135,000 PfSPZ/immunization
* Group 4: 4 or 6 doses of 135,000 PfSPZ/immunization.

If > 80% protective efficacy is not achieved in Groups 1, 2, or 3, volunteers in Group 4 will receive a fifth and sixth dose.

DETAILED DESCRIPTION:
The first clinical trial of the Pf SPZ vaccine is a Phase 1 trial in non-immune healthy adult volunteers. Sanaria is the Sponsor and PATH MVI is funding the trial. The study will be conducted as a collaborative effort between Sanaria, PATH MVI, the NMRC Malaria Program (U.S. Military Malaria Vaccine Program), and the Center for Vaccine Development at the University of Maryland at Baltimore (CVD-UMB). The study will take place at the NMRC Malaria Program Clinical Trials Center on the campus of the National Naval Medical Center in Bethesda, MD and at the CVD and/or General Clinical Research Center, UMB. The study is designed to evaluate the safety, tolerability, immunogenicity and protective efficacy of successively higher doses of the vaccine administered by the subcutaneous (SC) or intradermal (ID) route.

There will be 4 groups of volunteers with each group comprised of a subset of volunteers who receive the vaccine by the SC route and a subset who receive the vaccine by the ID route.

Groups 1-3: The first 3 groups will receive 3 ascending doses of vaccine administered as 4 SC or ID injections separated by 4 week intervals (7,500 PfSPZ/dose, 30,000 PfSPZ/dose, and 135,000 PfSPZ/dose respectively). Each of these groups will be challenged a minimum of 3 weeks after the final dose by exposure to A. stephensi mosquitoes infected with P. falciparum sporozoites. All 3 groups will be followed for safety until 48 weeks after the first immunization.

Group 4: Group 4 will start a minimum of 3 weeks after the first immunization of Group 3. If there is > 80% efficacy in one or more of the subsets of Groups 1, 2, or 3 (SC or ID), Group 4 volunteers will receive 4 immunizations (just like Group 3) but will not have experimental challenge; they will simply be followed for safety for 12 months after the first immunization. The FDA has requested that we follow a group of volunteers receiving the highest dose (135 PfSPZ/immunization) without challenge at 3 weeks. However, if there is NOT > 80% efficacy in one of more subsets of Groups 1, 2, or 3, after a 6 month observation period, Group 4 volunteers will receive two additional monthly immunizations (Immunizations #5 and #6) followed by challenge at approximately 3 weeks after the sixth immunization. All volunteers in Group 4 will be followed for safety until 52 weeks after the first immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (male or non-pregnant female) 18-50 years of age, inclusive.
2. Able and willing to participate for the duration of the study.
3. Able and willing to provide written (not proxy) informed consent.
4. Women of childbearing potential must agree to use effective means of birth control through the duration of the study.
5. Willing to refrain from blood donation (except as required in this study) for 3 years following P. falciparum challenge.
6. Agree not to travel to a malaria endemic region during the entire course of the trial.

Exclusion Criteria:

1. Any history of malaria infection, or travel to a malaria endemic region within 6 months prior to first immunization.
2. History of long term residence (>5 years) in area known to have significant transmission of P. falciparum.
3. Positive HIV, HBsAg or HCV serology. Positive sickle cell screening test.
4. Has evidence of increased cardiovascular disease risk (defined as > 10%, 5 year risk) as determined by the method of Gaziano (Gaziano 2008). Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/mm2), reported diabetes status, and blood pressure.
5. Current use of systemic immunosuppressant pharmacotherapy.
6. An abnormal EKG, defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
7. Current significant medical condition (cardiovascular, hepatic, renal, or hematological) or evidence of any other serious underlying medical condition identified by medical history, physical examination, or laboratory examination.
8. History of a splenectomy.
9. History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the volunteer's participation in the protocol or compromise the scientific objectives. This may include psychiatric disorders (such as personality disorders, anxiety disorders, or schizophrenia) or behavioral tendencies (including active alcohol or drug abuse) discovered during the screening process that in the opinion of the investigator would make compliance with the protocol difficult.
10. Plan for surgery between enrollment and challenge.
11. Females who are pregnant or nursing, females who plan on becoming pregnant or plan to nurse during the study period.
12. Known allergy to any component of the vaccine formulation, history of anaphylactic response to mosquito bites, retinal or visual field changes, or known allergy to the anti-malarial chloroquine phosphate, which will be used to treat volunteers developing malaria after P. falciparum challenge.
13. Participation in any study involving another investigational vaccine or drug within 90 days prior to the screening visit, or plan to participate in another investigational vaccine/drug research during or within 1 month following participation in this study.
14. Personal beliefs that prohibit the receiving of vaccine product containing human serum albumin within the diluent.
15. Use or planned use of any drug with anti-malarial activity that would coincide with immunization or challenge.
16. History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
17. Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone- proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of a non-replicating, metabolically active Plasmodium falciparum sporozoite (PfSPZ) vaccine in malaria-naïve healthy volunteers following multiple-dose subcutaneous (SC) or intradermal (ID) administration. | October 2010

SECONDARY OUTCOMES:
To evaluate PfSPZ vaccine-mediated protection against P. falciparum challenge in the 4 groups. | October 2010
To compare protective efficacy of the PfSPZ vaccine when given by SC versus ID administration in all groups. | October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Judith E Epstein, M.D., Principal Investigator — Naval Medical Research Center
Locations (2):
- United States (2):
  - The Center for Vaccine Development, University of Maryland (CVD/UMB), Baltimore, Maryland
  - Naval Medical Research Center (NMRC) Clinical Trials Center, on the campus of the National Naval Medical Center (NNMC), Bethesda, Maryland

REFERENCES:
- [Result] Epstein JE, Tewari K, Lyke KE, Sim BK, Billingsley PF, Laurens MB, Gunasekera A, Chakravarty S, James ER, Sedegah M, Richman A, Velmurugan S, Reyes S, Li M, Tucker K, Ahumada A, Ruben AJ, Li T, Stafford R, Eappen AG, Tamminga C, Bennett JW, Ockenhouse CF, Murphy JR, Komisar J, Thomas N, Loyevsky M, Birkett A, Plowe CV, Loucq C, Edelman R, Richie TL, Seder RA, Hoffman SL. Live attenuated malaria vaccine designed to protect through hepatic CD8(+) T cell immunity. Science. 2011 Oct 28;334(6055):475-80. doi: 10.1126/science.1211548. Epub 2011 Sep 8. PMID 21903775